CLINICAL TRIAL: NCT02055950
Title: A PROSPECTIVE STUDY TO COMPARE EARLY GRAFT FUNCTION OF RECIPIENTS OF SINGLE OR DUAL KIDNEY ORGANS STORED IN ICE COLD SOLUTION OR PULSED PERFUSION
Brief Title: Pulsed Perfusion for Marginal Kidneys
Acronym: PREDICTION
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICTION
Record Dates: First submitted 2014-01-28; First posted 2014-02-05 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney transplant; Marginal donors; Pulse perfusion; Graft function
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Kidney perfused by pulsatile machine
  Interventions: Procedure: Kidney perfused by pulsatile machine
- Kidney stored in refrigerated solution
  Interventions: Procedure: Storage of kidney in refrigerated solution

INTERVENTIONS:
Procedure: Storage of kidney in refrigerated solution
  Groups: Kidney stored in refrigerated solution
Procedure: Kidney perfused by pulsatile machine
  Groups: Kidney perfused by pulsatile machine

SUMMARY:
Trends in organ donor pool are characterized by an increasing age and a shift towards cerebrovascular diseases as primary causes of death. As a result, donors older than 60 years nowadays represent more than one fourth of the entire donor pool in Italy. This, along with an increasing number of patients on the waiting list for transplantation, prompted a growing use of organs from subjects older than 60 years that would have been considered unsuitable years ago. To improve graft outcomes, transplant of two older kidneys in the same recipient has been proposed. To optimize allocation of these organs to single or dual transplantation,a scoring system for kidneys, based on biopsy, with scores ranging from a minimum of 0 (indicating the absence of renal lesions) to a maximum of 12 (indicating the presence of marked changes in the renal parenchyma) has been suggested. According to this panel, kidneys with a score of 4 or lower are predicted to contain enough viable nephrons to be used as single transplants, those with a score of 5, 6, or 7 can be used as dual transplants, kidneys with a score greater than 7 are discarded. The survival of kidney grafts obtained from donors older than 60 years and allocated for single or dual transplantation on the basis of biopsy findings before transplantation was similar to that of single grafts from younger donors. To further improve these results, set-up of strategies to preserve organs is crucial to save the residual nephron mass and optimize outcomes of these marginal grafts. In this regard, over the past 30 years two methods of kidney preservation have been developed. With cold storage, the kidney is flushed once it is removed from the donor and placed in an ice-cooled container with preservation solution. With the use of pulsatile machine perfusion, the kidney is connected to a machine, which pumps a cold solution containing oxygen and nutrients through the kidney. This process allows for metabolism to continue in the kidney with end products being removed. The broad aim of the present study is to evaluate whether pulsatile machine perfusion of kidneys from older/marginal donors may provide better outcomes than static perfusion. To this purpose the outcome of recipients of perfused kidneys will be compared with the outcome of historical controls receiving non-perfused kidney selected and allocated on the basis of the same criteria and matched by gender, age and kidney histologic score.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 50 years or more and no more than 10 years older or younger than their corresponding donors;
* First single or double kidney transplant from deceased donors older than 60 years;
* Pre-implantation histologic evaluation and graft selection and allocation based on the histologic score and according to the Nord Italian Transplant (NIT) criteria;
* Written informed consent.

Exclusion Criteria:

* Any factor that according to the NIT selection criteria represent a contraindication to receive a deceased donor kidney transplant
* Need for specific de-sensitization protocols because of high immunological risk (according to NIT criteria) or participation in other concomitant intervention studies
* Vascular abnormalities/changes that preclude the possibility to perfuse the kidney grafts by a pulsatile machine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible to receive a single or dual transplant from older/marginal deceased donors identified according to the Nord Italia Transplant criteria who consent to receive perfused with a pulsatile machine.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) | 6 months after transplant.
Renal resistance | 6 hours after pulsatile machine perfusion
  Renal resistance is measured by graft ultrasound. It ranges from 0 to 1.

SECONDARY OUTCOMES:
Correlation between renal resistance measured at 6 hours after machine perfusion and renal histological score at pre-transplant biopsy | 6 hours after pulsatile machine perfusion
  The severity of changes in kidney at pre-transplant biopsy was quantified by a predefined histologic score. Changes in each evaluated component of the kidney tissue , vessels, glomeruli, tubules, and connective tissue, received a score ranging from 0 to 3. The sum of these scores was defined as the global kidney score, which could range from 0 to 12.
  Renal resistance is measured by graft ultrasound. It ranges from 0 to 1.
Correlation between renal resistances measured at 6 hours after pulsatile machine perfusion and intergraft resistances measured by ultrasound at 7 days and 6 months after transplant. | Changes from 7 days at 6 months after transplant .
  Renal resistances are measured by graft ultrasound. They range from 0 to 1.
Incidence of delayed graft function (DGF). | Within the first week after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cravedi, MD, Study Chair — IRCCS - Mario Negri Institute for Pharmacological Research; Giuseppe Remuzzi, MD, Principal Investigator — IRCCS - istituto di Ricerche Farmacologiche Mario Negri - A.O. Papa Giovanni XXIII BG; Giovanni Rota, MD, Principal Investigator — A.O. Papa Giovanni XXIII, Bergamo, Italy - U.O. Chirurgia Pediatrica; Salvatore De Pascale, MD, Principal Investigator — A.O. Papa Giovanni XXIII, Bergamo, Italy - U.O. Chirurgia Pediatrica; Francesco La Canna, MD, Principal Investigator — A.O. Papa Giovanni XXIII, Bergamo, Italy - U.O. Chirurgia Pediatrica; Giuseppe Piccolo, MD, Principal Investigator — NIT (North Italian Transplant); Giuseppe Rossini, MD, Principal Investigator — NIT (North Italian Transplant); Sergio Vesconi, MD, Principal Investigator — NIT (North Italian Transplant)
Locations (2):
- Italy (2):
  - A.O. Papa Giovanni XXIII - U.O. Nefrologia e Dialisi/U.O. Chirurgia Pediatrica, Bergamo
  - IRCCS Policlinico S.Matteo - UOS trapianto di Rene/U.O. Nefrologia, Pavia